CLINICAL TRIAL: NCT02162966
Title: Use Of High Dose Colistin in Multi Drug Resistant Gram Negative Infections in Critically Ill Adult Patients. Randomized Controlled Clinical Trial
Brief Title: Safety and Efficacy Study of High Dose Colistin
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: King Saud Medical City (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KSMC-CCD-AFM-002
Record Dates: First submitted 2014-05-21; First posted 2014-06-13 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Infectious Diseases
Keywords: colistin; ICU; critical care
MeSH Terms: conditions — Communicable Diseases | interventions — Colistin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Dose Colistin (Experimental): High dose colistin protocol
  Interventions: Drug: High Dose Colistin
- Standard Dose Colistin (Active Comparator): Standard dose of colistin
  Interventions: Drug: Standard Dose Colistin

INTERVENTIONS:
Drug: High Dose Colistin — High Dose Colistin
  Other Names: colistin
  Arms: High Dose Colistin
Drug: Standard Dose Colistin — Standard Dose Colistin
  Other Names: Colistin
  Arms: Standard Dose Colistin

SUMMARY:
Colistin is a rapidly acting bactericidal antimicrobial agent that possesses a post antibiotic effect against MDRO Gram-negative bacteria, such as as Pseudomonas aeruginosa, Acinetobacterbaumannii, and Klebsiella pneumonia.

ELIGIBILITY:
* Inclusion Criteria:

  1. Patient age more than or equal 18 years old.
  2. Patient has clinical signs and symptoms of infection with suspected or proven infection due to Carbapenem resistant microorganism.
  3. Patient was started with Empirical therapy of Colistin and positive MDRO within 5 days of empirical therapy.
* Exclusion Criteria:

  1. Patient age less than 18 years.
  2. Pregnant patient.
  3. If received Colistin treatment for less than 72 hours.
  4. Renal Replacement Therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2014-05; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Evaluate safety of high dose Colistin | 7 to 21 days after giving Colistin
  Evaluate the safety of high dose Colistin to treat MDRO infection in critically ill patients.
  The safety of high dose Colistin will be determined by number of participants whom renal function will be deviated from the baseline after administering high dose of Colistin.

SECONDARY OUTCOMES:
All cause mortality | 7 days after the end of therapy or at 28 days after enrollment
Ventilation free days | 28 days after enrollment
Length of ICU stay | 28 days after enrollment
Microbiological response | A day 7 and at the end of therapy
  whole body cultures will be done at day 7 of treatment and at the end of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed F Mady, PhD, Principal Investigator — King Saud Medical City
Locations (1):
- King Saud Medical City, Riyadh, Riyadh Region, Saudi Arabia